CLINICAL TRIAL: NCT00015275
Title: Pathophysiological Subtyping of Abnormalities in Cocaine Dependence
Brief Title: Pathophysiological Subtyping of Abnormalities in Cocaine Dependence - 9
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: New York MDRU (Other)
Masking: None | Purpose: Diagnostic
Other Study IDs: NIDA-5-0013-9; Y01-5-0013-9
Record Dates: First submitted 2001-04-18; First posted 2001-04-18 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2002-12

CONDITIONS: Cocaine-Related Disorders; Substance-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders

INTERVENTIONS:
Behavioral: Cocaine-Related Disorders

SUMMARY:
The purpose of this study is to define pathophysiological subtypes of abnormalities in subjects with cocaine dependence.

DETAILED DESCRIPTION:
The objective of this study is to define subgroups of patients with differential treatment outcome on the basis of differential baseline electrophysiological clusters.

ELIGIBILITY:
Inclusion Criteria:

Cocaine dependence. Seeking residential treatment.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0

PRIMARY OUTCOMES:
Identification of homogenous subgroups within total population of cocaine dependent adults

CONTACTS AND LOCATIONS:
Overall Officials: John Rotrosen, M.D., Principal Investigator — New York MDRU
Locations (1):
- New York MDRU, New York, New York, United States